CLINICAL TRIAL: NCT02081963
Title: A Randomized, Controlled Study of Combined Administration of Nebulized Amikacin in Patients With Acute Exacerbation of Non-Cystic Fibrosis Bronchiectasis
Brief Title: Combined Administration of Nebulized Amikacin in Patients With Acute Exacerbation of Non-Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qian Qi, assistant director, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCFB-AMK-01
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2015-11

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: Nebulized amikacin;; Non-Cystic Fibrosis Bronchiectasis;; Bacterial clearance rate of sputum；; Acute exacerbation.
MeSH Terms: interventions — Amikacin; Saline Solution

ARMS (2):
- Nebulized amikacin (Experimental): Participants receive nebulized amikacin BID for 14 days in combination with standard treatment.
  Interventions: Drug: Amikacin
- Nebulized normal saline (Other): Participants received nebulized normal saline BID for 14 days in combination with standard treatment.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Amikacin — Nebulized 0.2g of amikacin and 2 mL of normal saline twice a day for 14 days in combination with standard treatment.
  Arms: Nebulized amikacin
Drug: Normal saline — Nebulized 3 mL of normal saline twice a day for 14 days in combination with standard treatment.
  Arms: Nebulized normal saline

SUMMARY:
This is a multi-centered, randomized, controlled study to assess the efficacy, indications and adverse reactions of combined administration of nebulized amikacin in patients with acute exacerbation of non-cystic fibrosis bronchiectasis and to evaluate whether inhaled antibiotics are more likely to cause bacterial resistance.

DETAILED DESCRIPTION:
Objective: To assess the efficacy, indications and adverse reactions of combined administration of nebulized amikacin in patients with acute exacerbation of non-cystic fibrosis bronchiectasis and to evaluate whether inhaled antibiotics are more likely to cause bacterial resistance.

Methods: Patients with acute exacerbation of non-cystic fibrosis bronchiectasis will be randomly assigned to the observer group (participants receive nebulized amikacin BID for 14 days in combination with standard treatment) or the control group (participants receive nebulized 0.9% saline BID for 14 days in combination with standard treatment). The primary endpoint was bacterial clearance rate of sputum.

Expected results: Compared with the control group, bacterial clearance rate of sputum of the observer Group will increase significantly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female study subjects ≥18 years of age and ≤80 years of age;
* Confirmed diagnosis of idiopathic bronchiectasis or postinfectious bronchiectasis;
* Confirmation of infection with Pseudomonas aeruginosa at screening;
* Are sensitive to amikacin;
* Acute exacerbation of bronchiectasis.

Exclusion Criteria:

* Bronchiectasis due to special causes;
* Smokers;
* Are associated with bronchial asthma;
* Have any serious or active medical or psychiatric illness;
* Be allergic to amikacin or not tolerant to nebulised amikacin(FEV1 reduces ≥15% after inhaling amikacin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Li, Professor, Study Director — Director
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were screened and randomized at five tertiary hospitals in Shandong Province, China.
Pre-assignment Details: A total of 178 patients were screened in this study, and 26 unquali-fied patients (14.6%) were excluded.
Period: Overall Study
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Started | 79 | 73
Completed | 74 | 69
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline | Total
Number analyzed (Participants) | 79 | 73 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 67 | 137
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Nine patients were excluded from the final analysis due to dropout, 5 in the intervention group (6.3%) and 4 in the control group (5.6%).
  years
    number analyzed (Participants) | 74 | 69 | 143
    (all) | 57.3 (13.0) | 56.5 (10.8) | 56.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Nine patients were excluded from the final analysis due to dropout, 5 in the intervention group (6.3%) and 4 in the control group (5.6%).
  Participants
    number analyzed (Participants) | 74 | 69 | 143
    Female | 46 | 37 | 83
    Male | 28 | 32 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Nine patients were excluded from the final analysis due to dropout, 5 in the intervention group (6.3%) and 4 in the control group (5.6%).
  participants
    China: number analyzed (Participants) | 74 | 69 | 143
    China | 74 | 69 | 143

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Clearance Rate of Sputum
Description: The bacterial eradication rate of the sputum was calculated by the number of P. aeruginosa-eradicated cases according to sputum culture testing result. Sputum samples were collected in the morning after toothbrushing and gargling, before the patients used any medicine. Eligible sputum samples were defined as having ≥25 white blood cells/highpower field and ≤10 epithelial cells/high-power field; the samples were sent for testing within 60 min. Sputum samples were collected again after 14 days. If the second sputum culture test showed a negative result after the first one had been positive, it was defined as eradicated.
Time Frame: after 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Number analyzed (Participants) | 74 | 69
Participants | 38 | 16

2. Secondary Outcome: Total Sputum Weight (Collected Over 24 h) After 14 Days of Treatment
Time Frame: after 14 days
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Number analyzed (Participants) | 74 | 69
g | 18.4 (20.2) | 16.5 (20.8)

3. Secondary Outcome: Sputum Property Score After 14 Days of Treatment
Description: The sputum properties were graded from 1 to 4, with 1 being assigned to transparent mucous sputum, 2 to yellow purulent sputum, 3 to green purulent sputum, and 4 to black green purulent sputum. Higher scores mean a worse outcome.
Time Frame: after 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Number analyzed (Participants) | 74 | 69
score on a scale | 1.3 (0.6) | 1.3 (0.6)

4. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) (Percent of Predicted for Age) After 14 Days of Treatment
Time Frame: after 14 days
Measure: Mean (Standard Deviation); unit: Percent of Predicted
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Number analyzed (Participants) | 74 | 69
Percent of Predicted | 56.9 (23.9) | 60.0 (25.3)

5. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) After 14 Days of Treatment
Time Frame: after 14 days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
Number analyzed (Participants) | 74 | 69
L | 1.3 (0.7) | 1.5 (0.7)

ADVERSE EVENTS:
Arm/Group | Nebulized Amikacin | Nebulized Normal Saline
All-Cause Mortality (participants affected / at risk) | 1/79 | 1/73
Serious Adverse Events (participants affected / at risk) | 3/79 | 1/73
Other Adverse Events (participants affected / at risk) | 1/79 | 1/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebulized Amikacin (N=79) | Nebulized Normal Saline (N=73)
bronchospasms (Respiratory, thoracic and mediastinal disorders) | 2 | 1
nausea (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebulized Amikacin (N=79) | Nebulized Normal Saline (N=73)
nausea (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes